CLINICAL TRIAL: NCT02678715
Title: Effectiveness of Three Oral Devices as Mouthguard in Electroconvulsive Therapy.
Brief Title: Effectiveness of Three Oral Devices as Mouthguard in Electroconvulsive Therapy. Randomized Crossover Clinical Trial.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment period too long
Sponsor: Eva Willaert Jiménez-Pajarero (Other)
Responsible Party: Sponsor-Investigator, Eva Willaert Jiménez-Pajarero, DDS, PhD, University of Barcelona
Organization: University of Barcelona (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: AC089/15
Record Dates: First submitted 2016-01-25; First posted 2016-02-10 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Temporomandibular Joint Dysfunction Syndrome; Tooth Injuries; Dental Occlusion, Traumatic
MeSH Terms: conditions — Temporomandibular Joint Dysfunction Syndrome; Tooth Injuries; Dental Occlusion, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence SB-CA-SM (Experimental): Solubrux®+ Customized Appliance + Somatics®
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®
- Sequence SB-SM-CA (Experimental): Solubrux®+Somatics®+Customized Appliance
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®
- Sequence CA-SB-SM (Experimental): Customized Appliance+Solubrux®+Somatics®
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®
- Sequence CA-SM-SB (Experimental): Customized Appliance+Somatics®+Solubrux®
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®
- Sequence SM-SB-CA (Experimental): Somatics®+Solubrux®+Customized Appliance
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®
- Sequence SM-CA-SB (Experimental): Somatics®+ Customized Appliance+Solubrux®
  Interventions: Device: Solubrux®; Device: Customized Appliance; Device: Somatics®

INTERVENTIONS:
Device: Solubrux® — prefabricated device adaptable by temperature
Device: Customized Appliance — customized device fabricated in the dental laboratory
Device: Somatics® — standard device

SUMMARY:
This observer-blind crossover intervention study aims to determine the most effective type of device as oral mouthguard in modified-Electroconvulsive Therapy (m-ECT) comparing three types of devices: standard, prefabricated and manufactured in the dental laboratory.

Patients from the ECT Unit of Psychiatric Department of the University Hospital of Bellvitge will use the three devices at a random sequence during the twelve treatment sessions, so each device (A, B, C) will be used for two weeks, that is, for four consecutive sessions.

DETAILED DESCRIPTION:
Treatment with electroconvulsive therapy will involve the application of 12 m-ECT sessions at the rate of two sessions for six weeks according to the protocol established in the ECT Unit of the Department of Psychiatry at the University Hospital of Bellvitge.

Two devices, SB and CA, will be prepared for each patient and placed in mouth before anesthesia by one operator. This operator will assign a randomized sequence of use of the three devices (SB, CA or SM). Device SM will be the sole protector that will be placed after the anesthesia by nurse.

The outcome assessor will the scans pre- and post-session m-ECT and collect data, accede the surgery room before the session with the patient conscious and perform the exploration. This outcome assessor will leave the operating room during the procedure for the application of m-ECT an come back an hour later for the post-examination session.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have an intellectual level that allows a proper communication and must agree to cooperate in all tests and exams required by the study protocol.
* Obtaining written informed consent for participating in the project (model consent form)
* The patient must have enough teeth in the upper arch or being a carrier of a stable removable prosthesis.

Exclusion Criteria:

* Being in a maintenance ECT program.
* Receiving ECT during the six months prior to the index episode.
* Pregnancy and lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-02; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
temporomandibular pain | through study completion, an average of six weeks
  Continuous quantitative variable assessed by visual analogue scale (VAS) of 100 mm in length, marking the end as no pain (source) or the worst pain imaginable (final)

SECONDARY OUTCOMES:
Dental fractures | through study completion, an average of six weeks
  Dichotomic qualitative variable assessed by inspection: 0= 0 fractures; 1=≥1 fractures
Dental mobility assessed by Periotest® | through study completion, an average of six weeks
  Continuous quantitative /qualitative ordinal assessed by an electronic instrument that uses an ultrasonically vibrating probe (Periotest®) to assess dental mobility.
Oral soft tissues injuries | through study completion, an average of six weeks
  Dichotomic qualitative variable assessed by inspection: 0= 0 lesions; 1=≥1 lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided